# Brief Group Intervention Based on Acceptance and Commitment Therapy (ACT) for Problem Gambling: A Pilot Study

ID: 2025-81

Document date: February 23, 2025

Principal Investigators: Francisco Montesinos, Ph.D.- David Lobato, Ph.D.

**Study Protocol and Statistical Analysis Plan** 

# **Study Protocol**

# **Objective**

To examine the preliminary feasibility and acceptability of a brief group-based psychological intervention grounded in Acceptance and Commitment Therapy (ACT), aimed at young individuals exhibiting problematic gambling behaviors.

# Design

Open label pilot study

# **Methods**

After receiving detailed information about the structure and characteristics of the study, participants who provide written informed consent will undergo individual assessments to determine their eligibility. The assessment will include a structured interview and standardized questionnaires. Eligible participants will complete standardized questionnaires both before and after the intervention. The sample will consist of five participants who will receive an online group-based psychological treatment comprising eight weekly sessions, each lasting approximately 90 minutes.

## **Intervention Protocol**

#### Session 1: Introduction to ACT and Values Clarification

Through metaphors and experiential exercises, such as the "garden" metaphor, participants will explore meaningful life domains (e.g., family, relationships, health, education/work, leisure) that may have been overshadowed by gambling behavior.

# **Session 2: Acceptance and Cognitive Defusion**

Participants will be trained in cognitive defusion and acceptance strategies using exercises such as "the mind narrator," aimed at altering their relationship with automatic gambling-related thoughts.

#### **Session 3: Mindfulness**

Mindfulness practices focused on present-moment awareness, such as the "body scan" and "conscious breathing," will be introduced to help participants observe their thoughts, emotions, and bodily sensations without immediate reaction. This skill is expected to enhance recognition of gambling-related impulses and improve emotional regulation.

# **Session 4: Establishing the Observer Self Perspective**

The session will address how individuals identify with self-labels and narratives that foster hopelessness. Experiential exercises will be used to cultivate a more flexible and expansive perspective, reducing the influence of these narratives on behavior.

## **Session 5: Committed Action and Goal Setting**

Participants will work on identifying and formulating concrete personal goals aligned with their values. Strategies will be developed to support deliberate action toward these goals, even in the presence of emotional discomfort or gambling urges.

# Session 6: The Trap of Experiential Avoidance and Psychological Flexibility

The session will explore how gambling may serve as an escape from difficult emotions such as sadness, anxiety, or guilt. Through metaphors and experiential exercises, participants will be trained to remain in contact with these complex emotions without avoidance, thereby expanding their repertoire for coping with distress.

# **Session 7: Committed Action and Overcoming Barriers**

Internal and external barriers to value-consistent action—such as gambling urges, fear of failure, or aversive thoughts (e.g., "there's no point in trying," "I'm sure I can't do it")—will be identified. Practical exercises will be used to train flexible responses to these barriers.

## **Session 8: Consolidation and Maintenance Planning**

Key learnings will be reviewed, and an individualized action plan will be developed to sustain commitment to value-driven actions in the medium and long term. Potential risk situations that may trigger gambling urges will be identified, and coping strategies will be practiced.

# **Statistical Analysis Plan (SAP)**

Given the exploratory nature of the study and the small sample size, non-parametric tests will be employed to analyze the results (pre-, post-, and follow-up group mean comparisons). An analysis of variance will be conducted to determine the specific contribution of each independent variable and potential interactions among them. Additionally, the Jacobson and Truax (1991) method will be applied to estimate the clinical significance of the intervention effects.